CLINICAL TRIAL: NCT06178562
Title: Improving Clinical Outcomes in Infants With Pierre Robin Syndrome: A Randomized Controlled Study of Intermittent Oro-Esophageal Tube Feeding vs. Nasogastric Tube Feeding
Brief Title: Intermittent Oro-Esophageal Tube Feeding vs. Nasogastric Tube Feeding in Infants With Pierre Robin Syndrome
Acronym: PRS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: ethical issues
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Research Director, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-KY-0049-001
Record Dates: First submitted 2023-12-12; First posted 2023-12-21 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Pierre-Robin Syndrome; Dysphagia
Keywords: Infant; Pierre Robin Syndrome; Dysphagia; Rehabilitation
MeSH Terms: conditions — Pierre Robin Syndrome; Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outside of the research, all participating staff were required to avoid unnecessary contact with the patients enrolled and were instructed to strictly adhere to the confidentiality agreement regarding the study. The personnel responsible for data collection and assessment were not involved in other parts of the study and were unaware of the study design. Additionally, all assessments were conducted under the supervision of the principal investigator to ensure objectivity. All staff involved in the intervention underwent rigorous training to ensure that the implementation followed the protocol. Additionally, the principal investigator of the study regularly supervised the process of intervention to ensure compliance with the predetermined protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IOE group (Experimental): IOE groups were given systematic therapy according to the routine treatment plan for PRS for 4 weeks. The main intervention measures included: 1) non-invasive ventilator treatment, generally at least once every night and typically not exceeding continuous daily usage.; 2) attention to feeding and sleeping positions, with a recommended sleeping position of lateral recumbent and the head of the bed raised by 20-30°; 3) swallowing function training, such as tongue muscle stretching training, assisted anterior jaw protrusion training, lemon ice stimulation to the soft palate, pharyngeal wall, etc., generally 5 days per week, twice per day, 5-20 minutes each time; 4) pulmonary ultrashort wave therapy, generally at least 2-3 times a week, and not more than once a day; 5) physical therapy, such as intensive training for gross motor functions including lifting the head, turning over, sitting, crawling, standing, etc., generally 3-5 days per week, 1-2 times per day, 5-20 min each time.
  Interventions: Behavioral: systematic therapy; Device: IOE
- PNG group (Active Comparator): PNG groups were given systematic therapy according to the routine treatment plan for PRS for 4 weeks. The main intervention measures included: 1) non-invasive ventilator treatment, generally at least once every night and typically not exceeding continuous daily usage.; 2) attention to feeding and sleeping positions, with a recommended sleeping position of lateral recumbent and the head of the bed raised by 20-30°; 3) swallowing function training, such as tongue muscle stretching training, assisted anterior jaw protrusion training, lemon ice stimulation to the soft palate, pharyngeal wall, etc., generally 5 days per week, twice per day, 5-20 minutes each time; 4) pulmonary ultrashort wave therapy, generally at least 2-3 times a week, and not more than once a day; 5) physical therapy, such as intensive training for gross motor functions including lifting the head, turning over, sitting, crawling, standing, etc., generally 3-5 days per week, 1-2 times per day, 5-20 min each time.
  Interventions: Behavioral: systematic therapy; Device: PNG

INTERVENTIONS:
Behavioral: systematic therapy — Both groups were given systematic therapy according to the routine treatment plan for PRS for 4 weeks. The main intervention measures included: 1) non-invasive ventilator treatment, generally at least once every night and typically not exceeding continuous daily usage.; 2) attention to feeding and sleeping positions, with a recommended sleeping position of lateral recumbent and the head of the bed raised by 20-30°; 3) swallowing function training, such as tongue muscle stretching training, assisted anterior jaw protrusion training, lemon ice stimulation to the soft palate, pharyngeal wall, etc., generally 5 days per week, twice per day, 5-20 minutes each time; 4) pulmonary ultrashort wave therapy, generally at least 2-3 times a week, and not more than once a day; 5) physical therapy, such as intensive training for gross motor functions including lifting the head, turning over, sitting, crawling, standing, etc., generally 3-5 days per week, 1-2 times per day, 5-20 min each time.
Device: PNG — In PNG group, disposable gastric tubes were used for feeding to provide nutritional support. Each feeding was administered by a nurse using the infant's mother's breast milk through the tube. The amount of each feeding varied from 20 to 100 ml depending on the age of the infant, with feedings given every 2 to 3 hours, approximately 10 times per day. The duration of each feeding procedure ranged from 10 to 20 minutes. The total daily intake ranged from 200 to 1000 ml. Each tube was kept indwelling for 5 to 7 days. When the tube needed to be replaced, it was removed after the last feeding of a day and a new tube was to be inserted through the other nostril on the following morning to continue the nutritional support.
  Arms: PNG group
Device: IOE — The specific procedure was as follows: the infant was placed in a semi-recumbent or sitting position with the head fixed. Before each feeding, the infant's oral and nasal secretions were to be cleared. An intermittent oro-esophageal tube (Appendix) was appropriately lubricated with water on the head part. The professional medical staff held the tube and slowly inserted it through one side of the mouth into the upper part of the esophagus. The depth of insertion depended on the patient's age and height. After each feeding, the tube was immediately removed, and the patient was held upright for at least 30 minutes in case of reflux.
  Arms: IOE group

SUMMARY:
This was a randomized controlled study. The infants enrolled were randomly divided into the IOE group (with Intermittent Oro-Esophageal Tube Feeding, n=25) and the PNG group (with Nasogastric Tube Feeding, n=23), all receiving systemic therapy. Before and after 4-week treatment, pulmonary infection, swallowing function, nutritional status and body weight between the two group were compared.

DETAILED DESCRIPTION:
Pierre Robin Syndrome (PRS) can cause dysphagia. In China, persistent nasogastric tube feeding (PNG) is the mainstream choice as nutrition support in the dysphagic infants with PRS. However, PNG is associated with various complications, necessitating the exploration for a safer and more effective nutritional support approach. Therefore, this study aims to observe the clinical effect of intermittent oro-esophageal tube feeding (IOE) compared to PNG in the dysphagic infants with PRS who received systemic therapy.

This was a randomized controlled study. The infants enrolled were randomly divided into the IOE group (with IOE, n=25) and the PNG group (with PNG, n=23), all receiving systemic therapy. Before and after 4-week treatment, pulmonary infection, swallowing function, nutritional status and body weight between the two group were compared.

ELIGIBILITY:
Inclusion Criteria:

* meeting the diagnostic criteria for Pierre Robin sequence based on CT and X-ray examinations, combined with clinical manifestations and physical signs.
* with spontaneous vaginal birth, aged 1 to 12 months.
* with dysphagia screened by the water drinking test and further confirmed by the assessment of Dysphagia Disorders Survey (DDS), Dysphagia Severity Scale (DSS), or Schedule for Oral Motor Assessment (SOMA)
* before the treatment, the tube feeding was required and feasible after evaluation.
* stable vital signs.
* with nasogastric tubes placed before the treatment.
* sufficient human milk could be provided by the mothers of the patients (with the help of a manual suction device).

Exclusion Criteria:

* abnormalities in brain development or other neurological lesions revealed by CT or MRI scans.
* dysphagia caused by other diseases.
* other congenital malformations, such as Down syndrome, cleft lip, and palate, etc.
* severe systemic disease (such as severe infection, severe hepatic and renal dysfunction).
* participants who need to receive other therapy which would potentially affect the result of this study.

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients diagnosed as the pulmonary infection "Positive". | Day 1 and Day 28
  Once the symptoms of respiratory tract infection such as fever, cough, sputum, dyspnea, and respiratory distress were observed, the medical staffs would conduct the future exam. With the presence of rales on auscultation of both lungs, examination by CT, the routine blood test, and blood culture, the patients would be diagnosed as the pulmonary infection "Positive".

SECONDARY OUTCOMES:
Nutritional status-total protein | Day 1 and Day 28
  The relevant indicators include total protein (TP, g/L) from the blood test within 24h after admission and the last day of treatment, generally, with empty-stomach infants and in the morning.
Nutritional status-hemoglobin | Day 1 and Day 28
  The relevant indicators include hemoglobin (Hb, g/L)from the blood test within 24h after admission and the last day of treatment, generally, with empty-stomach infants and in the morning.
Nutritional status-albumin | Day 1 and Day 28
  The relevant indicators include albumin (ALB, g/L)from the blood test within 24h after admission and the last day of treatment, generally, with empty-stomach infants and in the morning.
Nutritional status-prealbumin | Day 1 and Day 28
  The relevant indicators include prealbumin (PA, mg/L) from the blood test within 24h after admission and the last day of treatment, generally, with empty-stomach infants and in the morning.
Body weight | Day 1 and Day 28
  Body weight measurement of the infants was conducted by the same nurse according to the relevant standards.
Swallowing function | Day 1 and Day 28
  The water drinking test (WDT) was used to assess the swallowing function due to the low feasibility of using swallowing imaging or flexible laryngoscopy in the infants with PRS and that these patients were unable to communicate and cooperate to complete the subjective components of most questionnaires. The patients were required to sit and drink 30 mL of warm water. Based on the completion of water intake and the occurrence of coughing, the results were divided into levels 1 to 6, with higher levels indicating a more severe degree of dysphagia.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Doctor, Study Chair — Site Coordinator of United Medical Group located in Miami
Locations (1):
- Zheng da yi fu yuan Hospital, Zhengzhou, China

IPD SHARING:
Plan to Share IPD: No